CLINICAL TRIAL: NCT04560010
Title: The Effect of Tranexamic Acid in Anticoagulated Patients Undergoing Total Shoulder Athroplasty
Brief Title: TXA in Anticoagulated Patients Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment rate was slower than anticipated
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00803
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Total Shoulder Athroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Subjects scheduled to undergo TSA (anatomic and reverse) will be randomized to receive one of two treatment options. This study will utilize a simple randomization approach to generate two-equal groups. All subjects have an equal chance (1:2) of getting randomized into one of the twp treatments groups: (1) Two doses of IV TXA, one before incision and the second 3 hours later. (2) control group - no TXA given. Randomization of each subject will be done on day of surgery. The randomization schedule will be generated using a computer software program such as randomization.com
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the anesthesiologist or surgeon will be blinded to the patient's group assignment, as they will be the one performing the treatment. All other stakeholders (patient, other caregivers, and research staff collecting the data) will be blinded to the patient's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid Injection (TXA) (Experimental): Subjects scheduled to undergo TSA (anatomic and reverse) will receive TXA before surgical incision and 3 hours later.
  Interventions: Drug: Tranexamic Acid Injection (TXA)
- No Tranexamic Acid Injection (TXA) given (No Intervention): Subjects scheduled to undergo TSA (anatomic and reverse) will receive no TXA.

INTERVENTIONS:
Drug: Tranexamic Acid Injection (TXA) — Injection of 1 gram of IV TXA before surgical plus 1 gram of IV TXA three hours later
  Arms: Tranexamic Acid Injection (TXA)

SUMMARY:
This is a randomized, single-blind, single-center study comparing calculated total blood loss, surgical drain output and hematoma formation in anticoagulated patients who receive 2 doses of Tranexamic Acid (TXA) versus control group undergoing anatomical and reverse total shoulder arthroplasty (TSA). Patients will be randomized to either receive 2 doses of IV TXA, first dose prior to surgical incision and second dose given 3 hours later or to the control group, where no TXA will be administered.

ELIGIBILITY:
Inclusion Criteria

* Patients older than 18 years old
* Patients undergoing scheduled primary anatomic total shoulder arthroplasty
* Patients undergoing scheduled primary reverse total shoulder arthroplasty
* Patients who consent to be randomized
* Preoperative use of anticoagulant or antiplatelet therapy within 10 days prior to surgery:

  * Coumadin (Warfarin)
  * Heparin
  * Low molecular weight heparin
  * Factor Xa inhibitors
  * Apixaban (Eliquis)
  * Rivarixaban (Xatelto)
  * Edoxaban (Savaysa)
  * Dabigatran (Pradaxa)
  * Clopidogrel (Plavix)
  * Prasugrel (Effient)
  * Ticagrelor (Brilinta)

Exclusion Criteria

* Patients younger than 18
* Patients who are pregnant* or breast-feeding women
* Patients who are allergic to tranexamic acid
* Patients scheduled for revision total shoulder arthroplasty
* Patients with proximal humerus fracture or fracture sequelae
* Patients who use estrogen containing medications (i.e. oral contraceptive pills)
* Patients who have acquired disturbances of color vision
* Patients with a history of any of the following diagnosis: '

  * Subarachnoid hemorrhage
  * Active intravascular clotting
  * Severe pulmonary disease (FEV <50% normal)
  * Plasma creatinine > 115 μmol/L in males, > 100 μmol/L in females, or hepatic failure)
  * (Renal impairment serum creatinine > 1.5 times the upper limit of normal NYU)
  * Preoperative anemia [Hemoglobin (Hb) < 11g/dL in females, Hb < 12 g/dL in males]
* Patients who refuse blood products
* Patients undergoing hormone replacement therapy
* Patients with diagnosed or self-reported cognitive dysfunction;
* Patients who are unable to understand or follow instructions;
* Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
* Patients with BMI over 50
* Any patient that the investigators feel cannot comply with all study related procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Hertling, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to the PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7.71) | 72 (6.944) | 72 (7.511)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Calculated Total Blood Loss
Description: "The volume of perioperative blood loss will be determined on the basis of the blood volume and change in hemoglobin from preoperatively to 1 day postoperatively. The volume of total perioperative blood loss will be determined according to the following formula:
  Total blood loss (ml) = 1000 x 〖Hb〗_loss/〖Hb〗_i"
Time Frame: Baseline to 24 hours post op
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Number analyzed (Participants) | 8 | 9
Milliliters | 0.6632 (0.2569) | 0.602 (0.2228)

2. Primary Outcome: Total Surgical Drain Output
Description: Surgical drain output will be recorded by floor nurse every 8 hours in EPIC. Data will be recorded up to 24 hours post-op if needed.
Time Frame: Up to 24 hours post-op
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Number analyzed (Participants) | 8 | 9
Milliliters | 131.3 (71.81) | 146.7 (75.7)

3. Secondary Outcome: Number of Participants With Presence of Hematoma
Description: Surgeon will assess for presence of hematoma at the 2-week follow up visit.
Time Frame: 2 weeks post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Number analyzed (Participants) | 8 | 9
Participants | 0 | 1

4. Secondary Outcome: Number of Participants Who Needed a Post-op Blood Transfusion
Time Frame: Up to 24 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

5. Secondary Outcome: Average Operative Time
Time Frame: During operation, up to 4 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Number analyzed (Participants) | 8 | 9
minutes | 88.25 (24.85) | 96 (19.33)

6. Secondary Outcome: Number of Patients Who Developed Adverse Events Such as Myocardial Infarction (MI), Pulmonary Embolus (PE), and/or Deep Vein Thrombosis (DVT)
Time Frame: Up until 30 days after last day of study participation, an average of 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Other (Not Including Serious) Adverse Events were collected for a period of 2 weeks. Serious Adverse Events and All-Cause Mortality was assessed up until 30 days after last day of study participation, up to 6 weeks
Arm/Group | Tranexamic Acid Injection (TXA) | No Tranexamic Acid Injection (TXA) Given
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04560010/Prot_SAP_001.pdf